CLINICAL TRIAL: NCT01956032
Title: Levodopa Carbidopa Intestinal Gel Home Titration Using Telemedicine: Evaluation of Use of Resources
Brief Title: Duodopa Home Titration Using Telemedicine: Evaluation of Use of Resources
Status: Completed | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P14-000
Record Dates: First submitted 2013-09-30; First posted 2013-10-08 (Estimated); Results first posted 2016-01-25 (Estimated); Last update posted 2016-02-23 (Estimated); Status verified 2016-01

CONDITIONS: Parkinson's Disease
Keywords: LCIG; Parkinson's disease; levodopa carbidopa intestinal gel; Telemedicine
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Participants with Parkinson's disease: Participants diagnosed with Parkinson's disease and have continued disabling motor complications despite optimized per-oral or other treatment regimens suitable for Duodopa treatment in accordance with the Swedish Summary of Products Characteristics.
  Other name for Duodopa is Levodopa Carbidopa Intestinal Gel (LCIG).

SUMMARY:
The purpose of this study was to evaluate the use of resources during titration of Duodopa at home.

DETAILED DESCRIPTION:
Telemedicine (TM) offers an alternative titration procedure allowing the start of Duodopa infusion at home. The study evaluated the use of resources, measured as the number of contacts and time spent by health care professionals (Duodopa nurse specialists and the study Investigators) and the TM technician, during Duodopa infusion at home. Data was collected from four (4) clinical centers in Sweden. Data collection period for each participant started at the decision to administer Duodopa treatment (Baseline) and ended when the Duodopa titration period was complete. Post-titration, the participants and caregiver were interviewed and the investigators and nurses answered a web based questionnaire on their experiences.

ELIGIBILITY:
Inclusion Criteria:

1. Suitable for Duodopa treatment in accordance with the Swedish Summary of Product Characteristics
2. Motivated and confident to test Duodopa home titration using TM
3. Participants who were able to handle the infusion pump and the TM equipment by themselves or with assistance, as determined by the Investigator
4. Understood and signed the study informed consent form

Exclusion Criteria:

1. Dementia or cognitive decline with Mini Mental State Examination score less than 24
2. Ongoing symptomatic depression, hallucinations or other psychotic behaviors without adequate treatment, as determined by the Investigator
3. Contraindications as described in the Swedish Summary of Product Characteristics: hypersensitivity to levodopa or carbidopa, narrow angle glaucoma, serious liver and kidney disease, severe heart failure, acute myocardial infarction, severe cardiac arrhythmias, recent or acute stroke, contraindications for adrenergic effects; pheochromocytoma, hyperthyroidism, cushing's syndrome, and other contraindications for abdominal surgery
4. Other reasons that made the participant unsuitable for home titration using TM, as determined by the Investigator

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with advanced Parkinson's disease admitted to movement disorder specialty clinics
Sampling Method: Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2013-09; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eva Dahl, MD, Study Director — AbbVie

REFERENCES:
- See also: Related Info — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Participants With Parkinson's Disease: Participants diagnosed with Parkinson's disease and have continued disabling motor complications despite optimized per-oral or other treatment regimens suitable for Duodopa treatment in accordance with the Swedish Summary of Products Characteristics.
Period: Overall Study
Arm/Group | Participants With Parkinson's Disease
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Participants With Parkinson's Disease
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65.5 (6.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 13

OUTCOME MEASURES:

1. Primary Outcome: Median Time Used by Investigator, Duodopa Nurse Specialist, Telemedicine (TM) Technician, and Participant
Description: Health care professional time was defined as the number of minutes the individual had contact with the participant visiting their home, assisting with TM equipment, or by telephone. TM technician time was defined as the number of minutes spent for setup, demounting, and adjustments to the TM equipment. Data are presented as the time in minutes for communication between the following individuals and summarized by the type of contact (all types, TM, telephone, home visit, and other): (1) Participant + Investigator time; (2) Participant + DNS time; (3) Participant + Investigator + DNS time; (4) Participant + TM technician time; (5) Total Investigator time; (6) Total DNS time; and (7) Total participant time.
Time Frame: From Baseline (Investigator's decision to start Duodopa treatment) until End of Titration (Investigator's decision to terminate Duodopa treatment) or up to approximately 14 days
Population: The analysis was performed using full analysis set (FAS), defined as all participants that started Duodopa titration.
Measure: Median (Full Range); unit: Minutes
Arm/Group | Participants With Parkinson's Disease
Number analyzed (Participants) | 15
Minutes
  Participant + Investigator: All Types (N=12) | 29.1 [3.0 to 39.0]
  Participant + Investigator: TM (N=12) | 22.2 [3.0 to 39.0]
  Participant + Investigator: Telephone (N=1) | 30.0 [30.0 to 30.0]
  Participant + Investigator: Home Visit (N=0) | NA [NA to NA] — Data were not available due to zero participants analyzed.
  Participant + Investigator: Other (N=0) | NA [NA to NA] — Data were not available due to zero participants analyzed.
  Participant + DNS: All Types | 317.4 [130.0 to 558.0]
  Participant + DNS: TM | 22.8 [10.0 to 97.0]
  Participant + DNS: Telephone (N=8) | 15.9 [1.0 to 46.0]
  Participant + DNS: Home Visit | 280.8 [75.0 to 437.0]
  Participant + DNS: Other (N=0) | NA [NA to NA] — Data were not available due to zero participants analyzed.
  Participant + Investigator + DNS: All Types | 45.0 [22.0 to 77.0]
  Participant + Investigator + DNS: TM | 42.0 [22.0 to 77.0]
  Participant + Investigator + DNS: Telephone (N=1) | 7.2 [7.2 to 7.2]
  Participant + Investigator + DNS: Home Visit (N=0) | NA [NA to NA] — Data were not available due to zero participants analyzed.
  Participant + Investigator + DNS: Other (N=0) | NA [NA to NA] — Data were not available due to zero participants analyzed.
  Participant + TM Technician: All Types | 100.2 [60.0 to 240.0]
  Participant + TM Technician: TM (N=1) | 1.8 [1.8 to 1.8]
  Participant + TM Technician: Telephone (N=1) | 4.2 [4.2 to 4.2]
  Participant + TM Technician: Home Visit | 100.2 [60.0 to 240.0]
  Participant + TM Technician: Other (N=0) | NA [NA to NA] — Data were not available due to zero participants analyzed.
  Total DNS: All Types | 349.2 [166.0 to 603.0]
  Total DNS: TM | 78.6 [41.0 to 132.0]
  Total DNS: Telephone (N=8) | 15.9 [1.0 to 50.0]
  Total DNS: Home Visit | 280.8 [75.0 to 437.0]
  Total DNS: Other (N=0) | NA [NA to NA] — Data were not available due to zero participants analyzed.
  Total Investigator: All Types | 73.8 [29.0 to 112.0]
  Total Investigator: TM | 57.0 [29.0 to 112.0]
  Total Investigator: Telephone (N=1) | 37.2 [37.2 to 37.2]
  Total Investigator: Home Visit (N=0) | NA [NA to NA] — Data were not available due to zero participants analyzed.
  Total Investigator: Other (N=0) | NA [NA to NA] — Data were not available due to zero participants analyzed.
  Total Participant: All Types | 532.8 [251.0 to 878.0]
  Total participant: TM | 100.2 [43.0 to 171.0]
  Total Participant: Telephone (N=8) | 15.9 [5.0 to 80.0]
  Total Participant: Home Visit | 345.0 [165.0 to 677.0]
  Total Participant: Other (N=0) | NA [NA to NA] — Data were not available due to zero participants analyzed.

2. Primary Outcome: Median Number of Contacts
Description: Contacts (total, TM, telephone, home visit, and other) during the study period between the participant, the health care professional (the DNS and the Investigator) and TM technician were counted and summarized by type. Data are presented as number of contacts per participant with a minimum and maximum range.
Time Frame: as for outcome 1
Population: The analysis was performed using FAS, defined as all participants that started Duodopa titration.
Measure: Median (Full Range); unit: Number of contacts
Arm/Group | Participants With Parkinson's Disease
Number analyzed (Participants) | 15
Number of contacts
  Total Contact With Participant: All Types | 19.0 [12.0 to 37.0]
  Total Contact With Participant: TM | 13.0 [7.0 to 23.0]
  Total Contact With Participant: Telephone | 1.0 [0.0 to 11.0]
  Total Contact With Participant: Home Visit | 5.0 [3.0 to 6.0]
  Total Contact With Participant: Other | 0.0 [0.0 to 0.0]
  Participant + Investigator: All Types | 3.0 [0.0 to 5.0]
  Participant + Investigator: TM | 2.0 [0.0 to 5.0]
  Participant + Investigator: Telephone | 0.0 [0.0 to 3.0]
  Participant + Investigator: Home Visit | 0.0 [0.0 to 0.0]
  Participant + Investigator: Other | 0.0 [0.0 to 0.0]
  Participant + DNS: All Types | 9.0 [5.0 to 22.0]
  Participant + DNS: TM | 5.0 [2.0 to 12.0]
  Participant + DNS: Telephone | 1.0 [0.0 to 7.0]
  Participant + DNS: Home Visit | 3.0 [1.0 to 4.0]
  Participant + DNS: Other | 0.0 [0.0 to 0.0]
  Participant + Investigator + DNS: All Types | 5.0 [2.0 to 11.0]
  Participant + Investigator + DNS: TM | 5.0 [2.0 to 11.0]
  Participant + Investigator + DNS: Telephone | 0.0 [0.0 to 1.0]
  Participant + Investigator + DNS: Home Visit | 0.0 [0.0 to 0.0]
  Participant + Investigator + DNS: Other | 0.0 [0.0 to 0.0]
  Participant + TM Technician: All Types | 2.0 [1.0 to 3.0]
  Participant + TM Technician: TM | 0.0 [0.0 to 1.0]
  Participant + TM Technician: Telephone | 0.0 [0.0 to 1.0]
  Participant + TM Technician: Home Visit | 2.0 [1.0 to 3.0]
  Participant + TM Technician: Other | 0.0 [0.0 to 0.0]

3. Secondary Outcome: Median Total Time for Titration
Description: The total time for titration period was defined as the number of minutes from the start of the pump after application of the naso-jejunal tube (Day 1) until Investigator's decision to terminate Duodopa treatment. Data are presented as time in minutes per participant with a minimum and maximum range.
Time Frame: From Day 1 (start of the pump after application of the naso-jejunal tube) until End of Titration (Investigator's decision to terminate Duodopa treatment) or up to approximately 14 days
Population: The analysis was performed using FAS, defined as all participants that started Duodopa titration.
Measure: Median (Full Range); unit: Minutes
Arm/Group | Participants With Parkinson's Disease
Number analyzed (Participants) | 15
Minutes | 4093.2 [2850.0 to 19925.0]

4. Secondary Outcome: Median Total Free Time of Participant
Description: Participant's daily free time was a maximum 24 hours, and was defined as the time spent on activities (e.g. work, household, chores, leisure time, travel, sleep, etc.) other than time spent on health care professional (the DNS and the Investigator) communication, dose adjustments and pump handling. Time for dose adjustments, health care professional communication via TM and pump handling were subtracted from the amount of participant's daily free time. The participant was asked to note the time used for independent dose adjustments and pump handling in a participant diary. Participant's total free time was calculated as the sum of participant's daily free time for all days during the titration period. Data are presented as time in minutes per participant with a minimum and maximum range.
Time Frame: as for outcome 3
Population: The analysis was performed using FAS, defined as all participants that started Duodopa titration.
Measure: Median (Full Range); unit: Minutes
Arm/Group | Participants With Parkinson's Disease
Number analyzed (Participants) | 15
Minutes | 3865.2 [2458.0 to 13659.0]

5. Secondary Outcome: Percentage of Participants Who Experienced Technical Events
Description: Technical events were defined as: any technical event; type A: TM equipment - mishandling; type B: TM equipment - intentional misuse; type C: TM equipment - technical problem; and type D: TM digital link. Technical problems were defined as: failure to answer video call, Intentional failure to answer video call, mechanical, electrical, failure to establish connection, interruptions, transmission quality, sound quality, image quality, and others. The percentage was calculated based on the number of participants in the FAS population.
Time Frame: as for outcome 1
Population: The analysis was performed using FAS, defined as all participants that started Duodopa titration.
Measure: Number; unit: Percentage of participants
Arm/Group | Participants With Parkinson's Disease
Number analyzed (Participants) | 15
Percentage of participants
  Any Technical Event | 73.3
  Type A: Failure to Answer Video Call | 13.3
  Type A: Other | 6.7
  Type B: Intentional Failure to Answer Video Call | 0.0
  Type B: Other | 0.0
  Type C: Mechanical | 13.3
  Type C: Electrical | 20.0
  Type C: Other | 33.3
  Type D: Failure to Establish Connection | 40.0
  Type D: Interruptions | 0.0
  Type D: Transmission Quality | 13.3
  Type D: Sound Quality | 33.3
  Type D: Image Quality | 6.7
  Type D: Other | 6.7

6. Secondary Outcome: Incidence of Technical Events Experienced by Participants
Description: Technical events were defined as: any technical event; type A: TM equipment - mishandling; type B: TM equipment - intentional misuse; type C: TM equipment - technical problem; and type D: TM digital link. Technical problems were defined as: failure to answer video call, Intentional failure to answer video call, mechanical, electrical, failure to establish connection, interruptions, transmission quality, sound quality, image quality, and others. The percentage was calculated based on the total number of technical events (34).
Time Frame: as for outcome 1
Population: The analysis was performed using FAS, defined as all participants that started Duodopa titration.
Measure: Number; unit: Percentage of technical events
Arm/Group | Participants With Parkinson's Disease
Number analyzed (Participants) | 15
Percentage of technical events
  Any Technical Event (N=11) | 100.0
  Type A: Failure to Answer Video Call (AVC) (N=2) | 5.9
  Type A: Other (N=1) | 2.9
  Type B: Intentional Failure to AVC (N=0) | NA — Data were not available due to zero participants analyzed.
  Type B: Other (N=0) | NA — Data were not available due to zero participants analyzed.
  Type C: Mechanical (N=2) | 8.8
  Type C: Electrical (N=3) | 14.7
  Type C: Other (N=5) | 14.7
  Type D: Failure to Establish Connection (N=6) | 32.4
  Type D: Interruptions (N=0) | NA — Data were not available due to zero participants analyzed.
  Type D: Transmission Quality (N=2) | 5.9
  Type D: Sound Quality (N=5) | 17.6
  Type D: Image Quality (N=1) | 2.9
  Type D: Other (N=1) | 2.9

7. Secondary Outcome: Percentage of Participants With Consequences
Description: Consequences due to technical events were defined as: any consequence, contact delay, re-establishment of connection, TM-call replaced by telephone call, failed scheduled contact, and other consequence. Data are summarized by type of technical event (type A: TM equipment - mishandling; type B: TM equipment - intentional misuse; type C: TM equipment - technical problem; and type D: TM digital link) and the percentage was calculated based on the number of participants in the FAS population.
Time Frame: as for outcome 1
Population: The analysis was performed using FAS, defined as all participants that started Duodopa titration.
Measure: Number; unit: Percentage of participants
Arm/Group | Participants With Parkinson's Disease
Number analyzed (Participants) | 15
Percentage of participants
  Any Consequence | 73.3
  Contact Delay: Type A | 6.7
  Contact Delay: Type B | 0.0
  Contact Delay: Type C | 20.0
  Contact Delay: Type D | 20.0
  Re-establishment of Connection: Type A | 6.7
  Re-establishment of Connection: Type B | 0.0
  Re-establishment of Connection: Type C | 26.7
  Re-establishment of Connection: Type D | 33.3
  TM-call Replaced by Telephone Call: Type A | 20.0
  TM-call Replaced by Telephone Call: Type B | 0.0
  TM-call Replaced by Telephone Call: Type C | 26.7
  TM-call Replaced by Telephone Call: Type D | 46.7
  Failed Scheduled Contact: Type A | 0.0
  Failed Scheduled Contact: Type B | 0.0
  Failed Scheduled Contact: Type C | 13.3
  Failed Scheduled Contact: Type D | 0.0
  Other Consequence: Type A | 0.0
  Other Consequence: Type B | 0.0
  Other Consequence: Type C | 13.3
  Other Consequence: Type D | 0.0

8. Secondary Outcome: Incidence of Consequences Due to Technical Events
Description: Consequences due to technical events were defined as: any consequence, contact delay, re-establishment of connection, TM-call replaced by telephone call, failed scheduled contact, and other consequence. Data are summarized by type of technical event (type A: TM equipment - mishandling; type B: TM equipment - intentional misuse; type C: TM equipment - technical problem; and type D: TM digital link) and the percentage was calculated based on the total number of consequences (43).
Time Frame: as for outcome 1
Population: The analysis was performed using FAS, defined as all participants that started Duodopa titration.
Measure: Number; unit: Percentage of consequences
Arm/Group | Participants With Parkinson's Disease
Number analyzed (Participants) | 15
Percentage of consequences
  Any Consequence (N=11) | 100.0
  Contact Delay: Type A (N=1) | 2.3
  Contact Delay: Type B (N=0) | NA — Data were not available due to zero participants analyzed.
  Contact Delay: Type C (N=3) | 7.0
  Contact Delay: Type D (N=3) | 11.6
  Re-establishment of Connection: Type A (N=1) | 2.3
  Re-establishment of Connection: Type B (N=0) | NA — Data were not available due to zero participants analyzed.
  Re-establishment of Connection: Type C (N=4) | 9.3
  Re-establishment of Connection: Type D (N=5) | 18.6
  TM-call Replaced by Telephone Call: Type A (N=3) | 7.0
  TM-call Replaced by Telephone Call: Type B (N=0) | NA — Data were not available due to zero participants analyzed.
  TM-call Replaced by Telephone Call: Type C (N=4) | 11.6
  TM-call Replaced by Telephone Call: Type D (N=7) | 23.3
  Failed Scheduled Contact: Type A (N=0) | NA — Data were not available due to zero participants analyzed.
  Failed Scheduled Contact: Type B (N=0) | NA — Data were not available due to zero participants analyzed.
  Failed Scheduled Contact: Type C (N=2) | 4.7
  Failed Scheduled Contact: Type D (N=0) | NA — Data were not available due to zero participants analyzed.
  Other Consequence: Type A (N=0) | NA — Data were not available due to zero participants analyzed.
  Other Consequence: Type B (N=0) | NA — Data were not available due to zero participants analyzed.
  Other Consequence: Type C (N=2) | 7.0
  Other Consequence: Type D (N=0) | NA — Data were not available due to zero participants analyzed.

9. Secondary Outcome: Percentage of Participants Who Experienced Technical Events, Summarized by Type of Consequence
Description: Technical events were defined as: any technical event; type A: TM equipment - mishandling; type B: TM equipment - intentional misuse; type C: TM equipment - technical problem; and type D: TM digital link). Data are summarized by type of consequence (contact delay, re-establishment of connection, TM-call replaced by telephone call, failed scheduled contact, and other consequence) and the percentage was calculated based on the number of participants in the FAS population.
Time Frame: as for outcome 1
Population: The analysis was performed using FAS, defined as all participants that started Duodopa titration.
Measure: Number; unit: Percentage of participants
Arm/Group | Participants With Parkinson's Disease
Number analyzed (Participants) | 15
Percentage of participants
  Any Technical Event | 73.3
  Type A: Contact Delay | 6.7
  Type A: Re-establishment of Connection | 6.7
  Type A: TM-call Replaced by Telephone Call | 20.0
  Type A: Failed Scheduled Contact Failure | 0.0
  Type A: Other Consequence | 0.0
  Type B: Contact Delay | 0.0
  Type B: Re-establishment of Connection | 0.0
  Type B: TM-call Replaced by Telephone Call | 0.0
  Type B: Failed Scheduled Contact Failure | 0.0
  Type B: Other Consequence | 0.0
  Type C: Contact Delay | 20.0
  Type C: Re-establishment of Connection | 26.7
  Type C: TM-call Replaced by Telephone Call | 26.7
  Type C: Failed Scheduled Contact Failure | 13.3
  Type C: Other Consequence | 13.3
  Type D: Contact Delay | 20.0
  Type D: Re-establishment of Connection | 33.3
  Type D: TM-call Replaced by Telephone Call | 46.7
  Type D: Failed Scheduled Contact Failure | 0.0
  Type D: Other Consequence | 0.0

10. Secondary Outcome: Incidence of Technical Events Experienced by Participants, Summarized by Type of Consequence
Description: Technical events were defined as: any technical event; type A: TM equipment - mishandling; type B: TM equipment - intentional misuse; type C: TM equipment - technical problem; and type D: TM digital link). Data are summarized by type of consequence (contact delay, re-establishment of connection, TM-call replaced by telephone call, failed scheduled contact, and other consequence) and the percentage was calculated based on the total number of technical events (34).
Time Frame: as for outcome 1
Population: The analysis was performed using FAS, defined as all participants that started Duodopa titration.
Measure: Number; unit: Percentage of technical events
Arm/Group | Participants With Parkinson's Disease
Number analyzed (Participants) | 15
Percentage of technical events
  Any Technical Event (N=11) | 100.0
  Type A: Contact Delay (N=1) | 2.9
  Type A: Re-establishment of Connection (N=1) | 2.9
  Type A: TM-call Replaced by Telephone Call (N=3) | 8.8
  Type A: Failed Scheduled Contact Failure (N=0) | NA — Data were not available due to zero participants analyzed.
  Type A: Other Consequence (N=0) | NA — Data were not available due to zero participants analyzed.
  Type B: Contact Delay (N=0) | NA — Data were not available due to zero participants analyzed.
  Type B: Re-establishment of Connection (N=0) | NA — Data were not available due to zero participants analyzed.
  Type B: TM-call Replaced by Telephone Call (N=0) | NA — Data were not available due to zero participants analyzed.
  Type B: Failed Scheduled Contact Failure (N=0) | NA — Data were not available due to zero participants analyzed.
  Type B: Other Consequence (N=0) | NA — Data were not available due to zero participants analyzed.
  Type C: Contact Delay (N=3) | 8.8
  Type C: Re-establishment of Connection (N=4) | 11.8
  Type C: TM-call Replaced by Telephone Call (N=4) | 14.7
  Type C: Failed Scheduled Contact Failure (N=2) | 5.9
  Type C: Other Consequence (N=2) | 8.8
  Type D: Contact Delay (N=3) | 14.7
  Type D: Re-establishment of Connection (N=5) | 23.5
  Type D: TM-call Replaced by Telephone Call (N=7) | 29.4
  Type D: Failed Scheduled Contact Failure (N=0) | NA — Data were not available due to zero participants analyzed.
  Type D: Other Consequence (N=0) | NA — Data were not available due to zero participants analyzed.

11. Secondary Outcome: Participant Experience of Duodopa Home Titration Using TM Assessed by Question Number 1: How Satisfied Were You With Using TM When Starting Duodopa?
Description: The experience of Duodopa home titration using TM was assessed using a sixteen item questionnaire via semi-structured interviews with the participant and caregiver (if applicable). The experience of Duodopa home titration using TM was measured by the participant on a scale from 1 to 7 for question number 1 (How satisfied were you with using TM when starting Duodopa?) where 1 was 'very dissatisfied' and 7 was 'very satisfied'. Data are presented as percentage of participants, calculated based on the number of participants in FAS with complete information.
Time Frame: as for outcome 1
Population: The analysis was performed using FAS with non-missing information.
Measure: Number; unit: Percentage of participants
Arm/Group | Participants With Parkinson's Disease
Number analyzed (Participants) | 14
Percentage of participants
  Scale 1 (Very Dissatisfied) | 0.0
  Scale 2 | 0.0
  Scale 3 | 0.0
  Scale 4 | 7.1
  Scale 5 | 7.1
  Scale 6 | 28.6
  Scale 7 (Very Satisfied) | 57.1

12. Secondary Outcome: Positive Participant Experience of Duodopa Home Titration Using TM Assessed by Question Number 2: Did You do Things When at Home That You Could Not Have Done if You Were Hospitalized During the Titration?
Description: The experience of Duodopa home titration using TM was assessed using a sixteen item questionnaire via semi-structured interviews with the participant and caregiver (if applicable). The experience of Duodopa home titration using TM was measured by the participant as 'yes' or 'no' for question number 2 (Did you do things when at home that you could not have done if you were hospitalized during the titration?) where 'yes' indicated a positive answer. Data are presented as percentage of participants with positive experience, calculated based on the number of participants in FAS with complete information.
Time Frame: as for outcome 1
Population: The analysis was performed using FAS with non-missing information.
Measure: Number; unit: Percentage of participants
Arm/Group | Participants With Parkinson's Disease
Number analyzed (Participants) | 14
Percentage of participants | 92.9

13. Secondary Outcome: Participant Experience of Duodopa Home Titration Using TM Assessed by Question Number 3: How Easy Was the TM Equipment to Use?
Description: The experience of Duodopa home titration using TM was assessed using a sixteen item questionnaire via semi-structured interviews with the participant and caregiver (if applicable). The experience of Duodopa home titration using TM was measured by the participant on a scale from 1 to 7 for question number 3 (How easy was the TM equipment to use?) where 1 was 'very hard' and 7 was 'very easy'. Data are presented as percentage of participants, calculated based on the number of participants in FAS with complete information.
Time Frame: as for outcome 1
Population: The analysis was performed using FAS with non-missing information.
Measure: Number; unit: Percentage of participants
Arm/Group | Participants With Parkinson's Disease
Number analyzed (Participants) | 14
Percentage of participants
  Scale 1 (Very Hard) | 0.0
  Scale 2 | 0.0
  Scale 3 | 0.0
  Scale 4 | 7.1
  Scale 5 | 7.1
  Scale 6 | 35.7
  Scale 7 (Very Easy) | 50.0

14. Secondary Outcome: Participant Experience of Duodopa Home Titration Using TM Assessed by Question Number 4: How Satisfied Were You With the Video Conversation With Your Investigator?
Description: The experience of Duodopa home titration using TM was assessed using a sixteen item questionnaire via semi-structured interviews with the participant and caregiver (if applicable). The experience of Duodopa home titration using TM was measured by the participant on a scale from 1 to 7 for question number 4 (How satisfied were you with the video conversation with your Investigator?) where 1 was 'very dissatisfied' and 7 was 'very satisfied'. Data are presented as percentage of participants, calculated based on the number of participants in FAS with complete information.
Time Frame: as for outcome 1
Population: The analysis was performed using FAS with non-missing information.
Measure: Number; unit: Percentage of participants
Arm/Group | Participants With Parkinson's Disease
Number analyzed (Participants) | 14
Percentage of participants
  Scale 1 (Very Dissatisfied) | 0.0
  Scale 2 | 0.0
  Scale 3 | 0.0
  Scale 4 | 0.0
  Scale 5 | 14.3
  Scale 6 | 28.6
  Scale 7 (Very Satisfied) | 57.1

15. Secondary Outcome: Participant Experience of Duodopa Home Titration Using TM Assessed by Question Number 5: How Satisfied Were You With the Video Conversation With Your DNS?
Description: The experience of Duodopa home titration using TM was assessed using a sixteen item questionnaire via semi-structured interviews with the participant and caregiver (if applicable). The experience of Duodopa home titration using TM was measured by the participant on a scale from 1 to 7 for question number 5 (How satisfied were you with the video conversation with your DNS?) where 1 was 'very dissatisfied' and 7 was 'very satisfied'. Data are presented as percentage of participants, calculated based on the number of participants in FAS with complete information.
Time Frame: as for outcome 1
Population: The analysis was performed using FAS with non-missing information.
Measure: Number; unit: Percentage of participants
Arm/Group | Participants With Parkinson's Disease
Number analyzed (Participants) | 14
Percentage of participants
  Scale 1 (Very Dissatisfied) | 0.0
  Scale 2 | 0.0
  Scale 3 | 0.0
  Scale 4 | 0.0
  Scale 5 | 7.1
  Scale 6 | 35.7
  Scale 7 (Very Satisfied) | 57.1

16. Secondary Outcome: Participant Experience of Duodopa Home Titration Using TM Assessed by Question Number 6: How Satisfied Were You With the 3-part Video Conversations (Both Investigator and DNS)?
Description: The experience of Duodopa home titration using TM was assessed using a sixteen item questionnaire via semi-structured interviews with the participant and caregiver (if applicable). The experience of Duodopa home titration using TM was measured by the participant on a scale from 1 to 7 for question number 6 (How satisfied were you with the 3-part video conversations with Investigator and DNS?) where 1 was 'very dissatisfied' and 7 was 'very satisfied'. Data are presented as percentage of participants, calculated based on the number of participants in FAS with complete information.
Time Frame: as for outcome 1
Population: The analysis was performed using FAS with non-missing information.
Measure: Number; unit: Percentage of participants
Arm/Group | Participants With Parkinson's Disease
Number analyzed (Participants) | 14
Percentage of participants
  Scale 1 (Very Dissatisfied) | 0.0
  Scale 2 | 0.0
  Scale 3 | 0.0
  Scale 4 | 0.0
  Scale 5 | 7.1
  Scale 6 | 21.4
  Scale 7 (Very Satisfied) | 71.4

17. Secondary Outcome: Participant Experience of Duodopa Home Titration Using TM Assessed by Question Number 7: How Satisfied Were You With the Amount of Time the DNS Were at Your Home?
Description: The experience of Duodopa home titration using TM was assessed using a sixteen item questionnaire via semi-structured interviews with the participant and caregiver (if applicable). The experience of Duodopa home titration using TM was measured by the participant on a scale from 1 to 7 for question number 7 (How satisfied were you with the amount of time the DNS were at your home?) where 1 was 'very dissatisfied' and 7 was 'very satisfied'. Data are presented as percentage of participants, calculated based on the number of participants in FAS with complete information.
Time Frame: as for outcome 1
Population: The analysis was performed using FAS with non-missing information.
Measure: Number; unit: Percentage of participants
Arm/Group | Participants With Parkinson's Disease
Number analyzed (Participants) | 14
Percentage of participants
  Scale 1 (Very Dissatisfied) | 0.0
  Scale 2 | 0.0
  Scale 3 | 0.0
  Scale 4 | 0.0
  Scale 5 | 7.1
  Scale 6 | 28.6
  Scale 7 (Very Satisfied) | 64.3

18. Secondary Outcome: Participant Experience of Duodopa Home Titration Using TM Assessed by Question Number 8: How Satisfied Were You With Having the Technical Equipment in Your Home?
Description: The experience of Duodopa home titration using TM was assessed using a sixteen item questionnaire via semi-structured interviews with the participant and caregiver (if applicable). The experience of Duodopa home titration using TM was measured by the participant on a scale from 1 to 7 for question number 8 (How satisfied were you with having the technical equipment in your home?) where 1 was 'very dissatisfied' and 7 was 'very satisfied'. Data are presented as percentage of participants, calculated based on the number of participants in FAS with complete information.
Time Frame: as for outcome 1
Population: The analysis was performed using FAS with non-missing information.
Measure: Number; unit: Percentage of participants
Arm/Group | Participants With Parkinson's Disease
Number analyzed (Participants) | 14
Percentage of participants
  Scale 1 (Very Dissatisfied) | 0.0
  Scale 2 | 0.0
  Scale 3 | 7.1
  Scale 4 | 0.0
  Scale 5 | 14.3
  Scale 6 | 0.0
  Scale 7 (Very Satisfied) | 78.6

19. Secondary Outcome: Participant Experience of Duodopa Home Titration Using TM Assessed by Question Number 9: How Satisfied Were You With the Technician's Visits to Set up and Dismantle the TM Equipment?
Description: The experience of Duodopa home titration using TM was assessed using a sixteen item questionnaire via semi-structured interviews with the participant and caregiver (if applicable). The experience of Duodopa home titration using TM was measured by the participant on a scale from 1 to 7 for question number 9 (How satisfied were you with the technician's visits to set up and dismantle the TM equipment?) where 1 was 'very dissatisfied' and 7 was 'very satisfied'. Data are presented as percentage of participants, calculated based on the number of participants in FAS with complete information.
Time Frame: as for outcome 1
Population: The analysis was performed using FAS with non-missing information.
Measure: Number; unit: Percentage of participants
Arm/Group | Participants With Parkinson's Disease
Number analyzed (Participants) | 14
Percentage of participants
  Scale 1 (Very Dissatisfied) | 0.0
  Scale 2 | 0.0
  Scale 3 | 7.1
  Scale 4 | 0.0
  Scale 5 | 7.1
  Scale 6 | 21.4
  Scale 7 (Very Satisfied) | 64.3

20. Secondary Outcome: Participant Experience of Duodopa Home Titration Using TM Assessed by Question Number 10: How Confident do You Feel Regarding the Pump and the Dose Adjustments?
Description: The experience of Duodopa home titration using TM was assessed using a sixteen item questionnaire via semi-structured interviews with the participant and caregiver (if applicable). The experience of Duodopa home titration using TM was measured by the participant on a scale from 1 to 7 for question number 10 (How confident do you feel regarding the pump and the dose adjustments?) where 1 was ' very unconfident' and 7 was 'very confident'. Data are presented as percentage of participants, calculated based on the number of participants in FAS with complete information.
Time Frame: as for outcome 1
Population: The analysis was performed using FAS with non-missing information.
Measure: Number; unit: Percentage of participants
Arm/Group | Participants With Parkinson's Disease
Number analyzed (Participants) | 14
Percentage of participants
  Scale 1 (Very Unconfident) | 0.0
  Scale 2 | 0.0
  Scale 3 | 0.0
  Scale 4 | 0.0
  Scale 5 | 14.3
  Scale 6 | 42.9
  Scale 7 (Very Confident) | 42.9

21. Secondary Outcome: Participant Experience of Duodopa Home Titration Using TM Assessed by Question Number 11: How Secure Did You Feel Being at Home and Communicating by TM, When Titrating Duodopa?
Description: The experience of Duodopa home titration using TM was assessed using a sixteen item questionnaire via semi-structured interviews with the participant and caregiver (if applicable). The experience of Duodopa home titration using TM was measured by the participant on a scale from 1 to 7 for question number 11 (How secure did you feel being at home and communicating by TM, when titrating Duodopa?) where 1 was 'very unsecure' and 7 was 'very secure'. Data are presented as percentage of participants, calculated based on the number of participants in FAS with complete information.
Time Frame: as for outcome 1
Population: The analysis was performed using FAS with non-missing information.
Measure: Number; unit: Percentage of participants
Arm/Group | Participants With Parkinson's Disease
Number analyzed (Participants) | 14
Percentage of participants
  Scale 1 (Very Unsecure) | 0.0
  Scale 2 | 0.0
  Scale 3 | 0.0
  Scale 4 | 7.1
  Scale 5 | 14.3
  Scale 6 | 14.3
  Scale 7 (Very Secure) | 64.3

22. Secondary Outcome: Positive Participant Experience of Duodopa Home Titration Using TM Assessed by Question Number 12: Knowing What You Know Now, Would You Rather Have Stayed in the Hospital to Start Duodopa Treatment?
Description: The experience of Duodopa home titration using TM was assessed using a sixteen item questionnaire via semi-structured interviews with the participant and caregiver (if applicable). The experience of Duodopa home titration using TM was measured by the participant as 'yes' or 'no' for question number 12 (Knowing what you know now, would you rather have stayed in the hospital to start Duodopa treatment?) where 'No' indicated a positive answer. Data are presented as percentage of participants with positive experience, calculated based on the number of participants in FAS with complete information.
Time Frame: as for outcome 1
Population: The analysis was performed using FAS with non-missing information.
Measure: Number; unit: Percentage of participants
Arm/Group | Participants With Parkinson's Disease
Number analyzed (Participants) | 14
Percentage of participants | 92.9

23. Secondary Outcome: Participant Experience of Duodopa Home Titration Using TM Assessed by Question Number 13 for Caregiver: How Satisfied Were You With the Titration at the Participant's Home?
Description: The experience of Duodopa home titration using TM was assessed using a sixteen item questionnaire via semi-structured interviews with the participant and caregiver (if applicable). The experience of Duodopa home titration using TM was measured by the caregiver on a scale from 1 to 7 for question number 13 (how satisfied were you with the titration at the participant's home?) where 1 was 'very dissatisfied' and 7 was 'very satisfied'. Data are presented as percentage of participants, calculated based on the number of participants in FAS with complete information.
Time Frame: as for outcome 1
Population: The analysis was performed using FAS with non-missing information.
Measure: Number; unit: Percentage of participants
Arm/Group | Participants With Parkinson's Disease
Number analyzed (Participants) | 9
Percentage of participants
  Scale 1 (Very Dissatisfied) | 0.0
  Scale 2 | 0.0
  Scale 3 | 0.0
  Scale 4 | 0.0
  Scale 5 | 0.0
  Scale 6 | 11.1
  Scale 7 (Very Satisfied) | 88.9

24. Secondary Outcome: Positive Participant Experience of Duodopa Home Titration Using TM Assessed by Question Number 14 for Caregiver: Where You Able to Perform Daily Activities During the Titration Period?
Description: The experience of Duodopa home titration using TM was assessed using a sixteen item questionnaire via semi-structured interviews with the participant and caregiver (if applicable). The experience of Duodopa home titration using TM was measured by the caregiver as 'yes' or 'no' for question number 14 (Where you able to perform daily activities during the titration period?) where 'yes' indicated a positive answer. Data are presented as percentage of participants with positive experience, calculated based on the number of participants in FAS with complete information.
Time Frame: as for outcome 1
Population: The analysis was performed using FAS with non-missing information.
Measure: Number; unit: Percentage of participants
Arm/Group | Participants With Parkinson's Disease
Number analyzed (Participants) | 9
Percentage of participants | 88.9

25. Secondary Outcome: Participant Experience of Duodopa Home Titration Using TM Assessed by Question Number 15 for Caregiver: How Confident Did You Feel About Helping With the Pump?
Description: The experience of Duodopa home titration using TM was assessed using a sixteen item questionnaire via semi-structured interviews with the participant and caregiver (if applicable). The experience of Duodopa home titration using TM was measured by the caregiver on a scale from 1 to 7 for question number 15 (How confident did you feel about helping with the pump?) where 1 was ' Very unconfident' and 7 was 'very confident'. Data are presented as percentage of participants, calculated based on the number of participants in FAS with complete information.
Time Frame: as for outcome 1
Population: The analysis was performed using FAS with non-missing information.
Measure: Number; unit: Percentage of participants
Arm/Group | Participants With Parkinson's Disease
Number analyzed (Participants) | 6
Percentage of participants
  Scale 1 (Very Unconfident) | 0.0
  Scale 2 | 0.0
  Scale 3 | 0.0
  Scale 4 | 0.0
  Scale 5 | 16.7
  Scale 6 | 16.7
  Scale 7 (Very Confident) | 66.7

26. Secondary Outcome: Positive Participant Experience of Duodopa Home Titration Using TM Assessed by Question Number 16 for Caregiver: Knowing What You Know Now, Would You Rather Have Had Your Spouse in the Hospital to Start Duodopa Treatment?
Description: From Baseline (Investigator's decision to start Duodopa treatment) until End of Titration (Investigator's decision to terminate Duodopa treatment) or up to approximately 14 days. The experience of Duodopa home titration using TM was measured by the caregiver as 'yes' or 'no' for question number 16 (knowing what you know now, would you rather have had your spouse in the hospital to start Duodopa treatment?) where 'No' indicated a positive answer. Data are presented as percentage of participants with positive experience, calculated based on the number of participants in FAS with complete information.
Time Frame: as for outcome 1
Population: The analysis was performed using FAS with non-missing information.
Measure: Number; unit: Percentage of participants
Arm/Group | Participants With Parkinson's Disease
Number analyzed (Participants) | 9
Percentage of participants | 100.0

27. Secondary Outcome: Investigator and DNS Experience of Duodopa Home Titration Using TM Assessed by Question Number 1: How Satisfied Were You With the TM Concept Comports With Your Clinical Needs?
Description: The experience of Duodopa home titration using TM was assessed using multiple web-based questionnaires by the Investigator and the DNS. The experience of Duodopa home titration using TM was measured on a scale from 1 to 7 for question number 1 (How satisfied were you with the TM concept comports with your clinical needs?) where 1 was 'very dissatisfied' and 7 was 'very satisfied'. Data are presented as percentage of participants, calculated based on the number of participants in FAS with complete information.
Time Frame: as for outcome 1
Population: The analysis was performed using FAS, defined as all participants that started Duodopa titration.
Measure: Number; unit: Percentage of participants
Arm/Group | Participants With Parkinson's Disease
Number analyzed (Participants) | 15
Percentage of participants
  Investigator Experience: Scale 1-Very Dissatisfied | 0.0
  Investigator Experience: Scale 2 | 0.0
  Investigator Experience: Scale 3 | 0.0
  Investigator Experience: Scale 4 | 6.7
  Investigator Experience: Scale 5 | 0.0
  Investigator Experience: Scale 6 | 53.3
  Investigator Experience: Scale 7-Very Satisfied | 40.0
  DNS Experience: Scale 1-Very Dissatisfied | 0.0
  DNS Experience: Scale 2 | 0.0
  DNS Experience: Scale 3 | 0.0
  DNS Experience: Scale 4 | 0.0
  DNS Experience: Scale 5 | 20.0
  DNS Experience: Scale 6 | 40.0
  DNS Experience: Scale 7-Very Satisfied | 40.0

28. Secondary Outcome: Investigator and DNS Experience of Duodopa Home Titration Using TM Assessed by Question Number 2: How Satisfied Were You With Using TM for Communication?
Description: The experience of Duodopa home titration using TM was assessed using multiple web-based questionnaires by the Investigator and the DNS. The experience of Duodopa home titration using TM was measured on a scale from 1 to 7 for question number 2 (How satisfied were you with using TM for communication?) where 1 was 'very dissatisfied' and 7 was 'very satisfied'. Data are presented as percentage of participants, calculated based on the number of participants in FAS with complete information.
Time Frame: as for outcome 1
Population: The analysis was performed using FAS, defined as all participants that started Duodopa titration.
Measure: Number; unit: Percentage of participants
Arm/Group | Participants With Parkinson's Disease
Number analyzed (Participants) | 15
Percentage of participants
  Investigator Experience: Scale 1-Very Dissatisfied | 0.0
  Investigator Experience: Scale 2 | 0.0
  Investigator Experience: Scale 3 | 0.0
  Investigator Experience: Scale 4 | 0.0
  Investigator Experience: Scale 5 | 13.3
  Investigator Experience: Scale 6 | 46.7
  Investigator Experience: Scale 7--Very Satisfied | 40.0
  DNS Experience: Scale 1-Very Dissatisfied | 0.0
  DNS Experience: Scale 2 | 0.0
  DNS Experience: Scale 3 | 0.0
  DNS Experience: Scale 4 | 6.7
  DNS Experience: Scale 5 | 0.0
  DNS Experience: Scale 6 | 46.7
  DNS Experience: Scale 7--Very Satisfied | 46.7

29. Secondary Outcome: Investigator and DNS Experience of Duodopa Home Titration Using TM Assessed by Question Number 3: How Satisfied Were You With Using TM for Clinical Assessments?
Description: The experience of Duodopa home titration using TM was assessed using multiple web-based questionnaires by the Investigator and the DNS. The experience of Duodopa home titration using TM was measured on a scale from 1 to 7 for question number 3 (How satisfied were you with using TM for clinical assessments?) where 1 was 'very dissatisfied' and 7 was 'very satisfied'. Data are presented as percentage of participants, calculated based on the number of participants in FAS with complete information.
Time Frame: as for outcome 1
Population: The analysis was performed using FAS, defined as all participants that started Duodopa titration.
Measure: Number; unit: Percentage of participants
Arm/Group | Participants With Parkinson's Disease
Number analyzed (Participants) | 15
Percentage of participants
  Investigator Experience: Scale 1-Very Dissatisfied | 0.0
  Investigator Experience: Scale 2 | 0.0
  Investigator Experience: Scale 3 | 6.7
  Investigator Experience: Scale 4 | 0.0
  Investigator Experience: Scale 5 | 6.7
  Investigator Experience: Scale 6 | 46.7
  Investigator Experience: Scale 7-Very Satisfied | 40.0
  DNS Experience: Scale 1-Very Dissatisfied | 0.0
  DNS Experience: Scale 2 | 0.0
  DNS Experience: Scale 3 | 0.0
  DNS Experience: Scale 4 | 6.7
  DNS Experience: Scale 5 | 13.3
  DNS Experience: Scale 6 | 40.0
  DNS Experience: Scale 7-Very Satisfied | 40.0

30. Secondary Outcome: Investigator and DNS Experience of Duodopa Home Titration Using TM Assessed by Question Number 4: How Satisfied Were You With the Image Quality for Your Assessment of the Participant?
Description: The experience of Duodopa home titration using TM was assessed using multiple web-based questionnaires by the Investigator and the DNS. The experience of Duodopa home titration using TM was measured on a scale from 1 to 7 for question number 4 (How satisfied were you with the image quality for your assessment of the participant?) where 1 was 'very dissatisfied' and 7 was 'very satisfied'. Data are presented as percentage of participants, calculated based on the number of participants in FAS with complete information.
Time Frame: as for outcome 1
Population: The analysis was performed using FAS, defined as all participants that started Duodopa titration.
Measure: Number; unit: Percentage of participants
Arm/Group | Participants With Parkinson's Disease
Number analyzed (Participants) | 15
Percentage of participants
  Investigator Experience: Scale 1-Very Dissatisfied | 0.0
  Investigator Experience: Scale 2 | 0.0
  Investigator Experience: Scale 3 | 6.7
  Investigator Experience: Scale 4 | 0.0
  Investigator Experience: Scale 5 | 0.0
  Investigator Experience: Scale 6 | 26.7
  Investigator Experience: Scale 7-Very Satisfied | 66.7
  DNS Experience: Scale 1-Very Dissatisfied | 0.0
  DNS Experience: Scale 2 | 0.0
  DNS Experience: Scale 3 | 0.0
  DNS Experience: Scale 4 | 0.0
  DNS Experience: Scale 5 | 20.0
  DNS Experience: Scale 6 | 33.3
  DNS Experience: Scale 7-Very Satisfied | 46.7

31. Secondary Outcome: Investigator and DNS Experience of Duodopa Home Titration Using TM Assessed by Question Number 5: How Satisfied Were You With the Sound Quality for Your Assessment of the Participant?
Description: The experience of Duodopa home titration using TM was assessed using multiple web-based questionnaires by the Investigator and the DNS. The experience of Duodopa home titration using TM was measured on a scale from 1 to 7 for question number 5 (How satisfied were you with the sound quality for your assessment of the participant?) where 1 was 'very dissatisfied' and 7 was 'very satisfied'. Data are presented as percentage of participants, calculated based on the number of participants in FAS with complete information.
Time Frame: as for outcome 1
Population: The analysis was performed using FAS, defined as all participants that started Duodopa titration.
Measure: Number; unit: Percentage of participants
Arm/Group | Participants With Parkinson's Disease
Number analyzed (Participants) | 15
Percentage of participants
  Investigator Experience: Scale 1-Very Dissatisfied | 0.0
  Investigator Experience: Scale 2 | 0.0
  Investigator Experience: Scale 3 | 6.7
  Investigator Experience: Scale 4 | 6.7
  Investigator Experience: Scale 5 | 26.7
  Investigator Experience: Scale 6 | 46.7
  Investigator Experience: Scale 7-Very Satisfied | 13.3
  DNS Experience: Scale 1-Very Dissatisfied | 0.0
  DNS Experience: Scale 2 | 0.0
  DNS Experience: Scale 3 | 0.0
  DNS Experience: Scale 4 | 13.3
  DNS Experience: Scale 5 | 26.7
  DNS Experience: Scale 6 | 40.0
  DNS Experience: Scale 7-Very Satisfied | 20.0

32. Secondary Outcome: Investigator and DNS Experience of Duodopa Home Titration Using TM Assessed by Question Number 6: How Satisfied Were You With the User Interphase for the TM Equipment?
Description: The experience of Duodopa home titration using TM was assessed using multiple web-based questionnaires by the Investigator and the DNS. The experience of Duodopa home titration using TM was measured on a scale from 1 to 7 for question number 6 (How satisfied were you with the user interphase for the TM equipment?) where 1 was 'very dissatisfied' and 7 was 'very satisfied'. Data are presented as percentage of participants, calculated based on the number of participants in FAS with complete information.
Time Frame: as for outcome 1
Population: The analysis was performed using FAS, defined as all participants that started Duodopa titration.
Measure: Number; unit: Percentage of participants
Arm/Group | Participants With Parkinson's Disease
Number analyzed (Participants) | 15
Percentage of participants
  Investigator Experience: Scale 1-Very Dissatisfied | 0.0
  Investigator Experience: Scale 2 | 0.0
  Investigator Experience: Scale 3 | 0.0
  Investigator Experience: Scale 4 | 0.0
  Investigator Experience: Scale 5 | 13.3
  Investigator Experience: Scale 6 | 13.3
  Investigator Experience: Scale 7-Very Satisfied | 73.3
  DNS Experience: Scale 1-Very Dissatisfied | 0.0
  DNS Experience: Scale 2 | 0.0
  DNS Experience: Scale 3 | 0.0
  DNS Experience: Scale 4 | 0.0
  DNS Experience: Scale 5 | 13.3
  DNS Experience: Scale 6 | 6.7
  DNS Experience: Scale 7-Very Satisfied | 80.0

33. Secondary Outcome: Investigator and DNS Experience of Duodopa Home Titration Using TM Assessed by Question Number 7: How Satisfied Were You With the Setup and Maintenance of the TM Equipment?
Description: The experience of Duodopa home titration using TM was assessed using multiple web-based questionnaires by the Investigator and the DNS. The experience of Duodopa home titration using TM was measured on a scale from 1 to 7 for question number 7 (How satisfied were you with the setup and maintenance of the TM equipment?) where 1 was 'very dissatisfied' and 7 was 'very satisfied'. Data are presented as percentage of participants, calculated based on the number of participants in FAS with complete information.
Time Frame: as for outcome 1
Population: The analysis was performed using FAS, defined as all participants that started Duodopa titration.
Measure: Number; unit: Percentage of participants
Arm/Group | Participants With Parkinson's Disease
Number analyzed (Participants) | 15
Percentage of participants
  Investigator Experience: Scale 1-Very Dissatisfied | 0.0
  Investigator Experience: Scale 2 | 0.0
  Investigator Experience: Scale 3 | 0.0
  Investigator Experience: Scale 4 | 0.0
  Investigator Experience: Scale 5 | 20.0
  Investigator Experience: Scale 6 | 60.0
  Investigator Experience: Scale 7-Very Satisfied | 20.0
  DNS Experience: Scale 1-Very Dissatisfied | 0.0
  DNS Experience: Scale 2 | 6.7
  DNS Experience: Scale 3 | 0.0
  DNS Experience: Scale 4 | 0.0
  DNS Experience: Scale 5 | 26.7
  DNS Experience: Scale 6 | 20.0
  DNS Experience: Scale 7-Very Satisfied | 46.7

34. Secondary Outcome: Investigator and DNS Experience of Duodopa Home Titration Using TM Assessed by Question Number 8: How Satisfied Were You Regarding Participant Safety Using TM?
Description: The experience of Duodopa home titration using TM was assessed using multiple web-based questionnaires by the Investigator and the DNS. The experience of Duodopa home titration using TM was measured on a scale from 1 to 7 for question number 8 (How satisfied were you regarding participant safety using TM?) where 1 was 'very dissatisfied' and 7 was 'very satisfied'. Data are presented as percentage of participants, calculated based on the number of participants in FAS with complete information.
Time Frame: as for outcome 1
Population: The analysis was performed using FAS, defined as all participants that started Duodopa titration.
Measure: Number; unit: Percentage of participants
Arm/Group | Participants With Parkinson's Disease
Number analyzed (Participants) | 15
Percentage of participants
  Investigator Experience: Scale 1-Very Dissatisfied | 0.0
  Investigator Experience: Scale 2 | 0.0
  Investigator Experience: Scale 3 | 0.0
  Investigator Experience: Scale 4 | 0.0
  Investigator Experience: Scale 5 | 13.3
  Investigator Experience: Scale 6 | 46.7
  Investigator Experience: Scale 7-Very Satisfied | 40.0
  DNS Experience: Scale 1-Very Dissatisfied | 0.0
  DNS Experience: Scale 2 | 0.0
  DNS Experience: Scale 3 | 6.7
  DNS Experience: Scale 4 | 0.0
  DNS Experience: Scale 5 | 6.7
  DNS Experience: Scale 6 | 20.0
  DNS Experience: Scale 7-Very Satisfied | 66.7

35. Secondary Outcome: Investigator and DNS Experience of Duodopa Home Titration Using TM Assessed by Question Number 9: How Satisfied Were You With the Participant Contact When Using TM?
Description: The experience of Duodopa home titration using TM was assessed using multiple web-based questionnaires by the Investigator and the DNS. The experience of Duodopa home titration using TM was measured on a scale from 1 to 7 for question number 9 (How satisfied were you with the participant contact when using TM?) where 1 was 'very dissatisfied' and 7 was 'very satisfied'. Data are presented as percentage of participants, calculated based on the number of participants in FAS with complete information.
Time Frame: as for outcome 1
Population: The analysis was performed using FAS, defined as all participants that started Duodopa titration.
Measure: Number; unit: Percentage of participants
Arm/Group | Participants With Parkinson's Disease
Number analyzed (Participants) | 15
Percentage of participants
  Investigator Experience: Scale 1-Very Dissatisfied | 0.0
  Investigator Experience: Scale 2 | 0.0
  Investigator Experience: Scale 3 | 0.0
  Investigator Experience: Scale 4 | 0.0
  Investigator Experience: Scale 5 | 6.7
  Investigator Experience: Scale 6 | 26.7
  Investigator Experience: Scale 7-Very Satisfied | 66.7
  DNS Experience: Scale 1-Very Dissatisfied | 0.0
  DNS Experience: Scale 2 | 0.0
  DNS Experience: Scale 3 | 0.0
  DNS Experience: Scale 4 | 6.7
  DNS Experience: Scale 5 | 6.7
  DNS Experience: Scale 6 | 20.0
  DNS Experience: Scale 7-Very Satisfied | 66.7

36. Secondary Outcome: Positive (Investigator and DNS) Experience of Duodopa Home Titration Using TM Assessed by Question Number 10: Did You Lack Any Dimensions in the Assessment of the Participant Using TM That You Have in the Classical Titration at Hospital?
Description: The experience of Duodopa home titration using TM was assessed using multiple web-based questionnaires by the Investigator and the DNS. The experience of Duodopa home titration using TM was measured as 'yes' or 'no' for question number 10 (Did you lack any dimensions in the assessment of the participant using TM that you have in the classical titration at hospital?) where 'No' indicated a positive answer. Data are presented as percentage of participants with positive experience, calculated based on the number of participants in FAS with complete information.
Time Frame: as for outcome 1
Population: The analysis was performed using FAS, defined as all participants that started Duodopa titration.
Measure: Number; unit: Percentage of participants
Arm/Group | Participants With Parkinson's Disease
Number analyzed (Participants) | 15
Percentage of participants
  Investigator Experience | 73.3
  DNS Experience | 60.0

37. Secondary Outcome: Investigator and DNS Experience of Duodopa Home Titration Using TM Assessed by Question Number 11: Compared to Classic Titration at Hospital - How Much Time Did You Spend on TM Communication Based on Real Communication Time for Participant Contact?
Description: The experience of Duodopa home titration using TM was assessed using multiple web-based questionnaires by the Investigator and the DNS. The experience of Duodopa home titration using TM was measured as 'more', 'equal' or 'less' for question number 11 (Compared to classic titration at hospital - how much time did you spend on TM communication based on real communication time for participant contact?) where 'more' indicated the most negative answer and 'less' indicated the most positive answer. Data are presented as percentage of participants, calculated based on the number of participants in FAS with complete information.
Time Frame: as for outcome 1
Population: The analysis was performed using FAS, defined as all participants that started Duodopa titration.
Measure: Number; unit: Percentage of participants
Arm/Group | Participants With Parkinson's Disease
Number analyzed (Participants) | 15
Percentage of participants
  Investigator Experience: More | 0.0
  Investigator Experience: Equal | 40.0
  Investigator Experience: Less | 60.0
  DNS Experience: More | 0.0
  DNS Experience: Equal | 6.7
  DNS Experience: Less | 93.3

38. Secondary Outcome: Investigator and DNS Experience of Duodopa Home Titration Using TM Assessed by Question Number 12: Compared to Classic Titration at Hospital - How Much Time Did You Spend on TM Communication Based on Booked Communication Time for Participant Contact?
Description: The experience of Duodopa home titration using TM was assessed using multiple web-based questionnaires by the Investigator and the DNS. The experience of Duodopa home titration using TM was measured as 'more', 'equal' or 'less' for question number 12 (Compared to classic titration at hospital - how much time did you spend on TM communication based on booked communication time for participant contact?) where 'more' indicated the most negative answer and 'less' indicated the most positive answer. Data are presented as percentage of participants, calculated based on the number of participants in FAS with complete information.
Time Frame: as for outcome 1
Population: The analysis was performed using FAS, defined as all participants that started Duodopa titration.
Measure: Number; unit: Percentage of participants
Arm/Group | Participants With Parkinson's Disease
Number analyzed (Participants) | 15
Percentage of participants
  Investigator Experience: More | 6.7
  Investigator Experience: Equal | 26.7
  Investigator Experience: Less | 66.7
  DNS Experience: More | 26.7
  DNS Experience: Equal | 13.3
  DNS Experience: Less | 60.0

39. Secondary Outcome: Investigator and DNS Experience of Duodopa Home Titration Using TM Assessed by Question Number 13: Compared to Classic Titration at Hospital - How Much Time Did You Spend on TM Communication Based on Time for Other Tasks Between Contacts?
Description: The experience of Duodopa home titration using TM was assessed using multiple web-based questionnaires by the Investigator and the DNS. The experience of Duodopa home titration using TM was measured as 'more', 'equal' or 'less' for question number 13 (Compared to classic titration at hospital - how much time did you spend on TM communication based on time for other tasks between contacts?) where 'more' indicated the most negative answer and 'less' indicated the most positive answer. Data are presented as percentage of participants, calculated based on the number of participants in FAS with complete information.
Time Frame: as for outcome 1
Population: The analysis was performed using FAS, defined as all participants that started Duodopa titration.
Measure: Number; unit: Percentage of participants
Arm/Group | Participants With Parkinson's Disease
Number analyzed (Participants) | 15
Percentage of participants
  Investigator Experience: More | 53.3
  Investigator Experience: Equal | 40.0
  Investigator Experience: Less | 6.7
  DNS Experience: More | 93.3
  DNS Experience: Equal | 6.7
  DNS Experience: Less | 0.0

40. Secondary Outcome: DNS Experience of Duodopa Home Titration Using TM Assessed by Question Number 14: How Satisfied Were You With Replacing the Participant Home Visit With TM Communication?
Description: The experience of Duodopa home titration using TM was assessed using multiple web-based questionnaires by the DNS. The experience of Duodopa home titration using TM was measured on a scale from 1 to 7 for question number 14 (How satisfied were you with replacing the participant home visit with TM communication?) where 1 was 'very dissatisfied' and 7 was 'very satisfied'. Data are presented as percentage of participants, calculated based on the number of participants in FAS with complete information.
Time Frame: as for outcome 1
Population: The analysis was performed using FAS, defined as all participants that started Duodopa titration.
Measure: Number; unit: Percentage of participants
Arm/Group | Participants With Parkinson's Disease
Number analyzed (Participants) | 15
Percentage of participants
  Scale 1 (Very Dissatisfied) | 0.0
  Scale 2 | 0.0
  Scale 3 | 0.0
  Scale 4 | 6.7
  Scale 5 | 13.3
  Scale 6 | 20.0
  Scale 7 (Very Satisfied) | 60.0

41. Secondary Outcome: Percentage of Participants With Clinical Global Impression - Improvement (CGI-I) in Parkinson's Disease Symptoms
Description: CGI-I was used to document the Investigator's impression of the participant's improvement in Parkinson's Disease symptoms throughout the study. The CGI-I was measured on a 7-point scale: 1=Very much improved; 2=Much improved; 3=Minimally improved; 4=No change; 5=Minimally worse; 6=Much worse; and 7=Very much worse, where 1 through 3 indicated positive answers. Data are presented as percentage of participants, calculated based on the number of participants in FAS with complete information.
Time Frame: as for outcome 1
Population: The analysis was performed using FAS with non-missing information.
Measure: Number; unit: Percentage of participants
Arm/Group | Participants With Parkinson's Disease
Number analyzed (Participants) | 14
Percentage of participants
  Very Much Improved | 28.6
  Much Improved | 71.4
  Minimally Improved | 0.0
  No Change | 0.0
  Minimally Worse | 0.0
  Much Worse | 0.0
  Very Much Worse | 0.0

42. Secondary Outcome: Number of Participants With Health Care Utilization Outside the TM Care Chain, Summarized by Type of Health Care Provider
Description: The number of participants with health care utilization outside the TM care chain was assessed and summarized by type of health care provider (general practitioner, emergency ward, other neurologist, and other).
Time Frame: as for outcome 1
Population: The analysis was performed using FAS, defined as all participants that started Duodopa titration.
Measure: Number; unit: Number of participants
Arm/Group | Participants With Parkinson's Disease
Number analyzed (Participants) | 15
Number of participants
  General Practitioner | 0
  Emergency Ward | 0
  Other Neurologist | 0
  Other | 1

43. Secondary Outcome: Number of Participants With Health Care Utilization Outside the TM Care Chain, Summarized by Type of Contact
Description: The number of participants with health care utilization outside the TM care chain was assessed and summarized by type of contact (other, telephone, home or outpatient visit, and hospitalization).
Time Frame: as for outcome 1
Population: The analysis was performed using FAS, defined as all participants that started Duodopa titration.
Measure: Number; unit: Number of participants
Arm/Group | Participants With Parkinson's Disease
Number analyzed (Participants) | 15
Number of participants
  Other | 0
  Telephone | 0
  Home or Outpatient Visit | 1
  Hospitalization | 0

44. Secondary Outcome: Median Time Spent for Health Care Utilization Outside the TM Care Chain
Description: The time spent in minutes for health care utilization outside the TM care chain was assessed. Data are presented as time in minutes with a minimum and maximum range.
Time Frame: as for outcome 1
Population: The analysis was performed using FAS with non-missing information.
Measure: Median (Full Range); unit: Minutes
Arm/Group | Participants With Parkinson's Disease
Number analyzed (Participants) | 1
Minutes | 190.8 [190.8 to 190.8]

ADVERSE EVENTS:
Time Frame: From signing of informed consent until 30 days or 5 half-lives from the last dose of Duodopa treatment or up to approximately 45 days
Description: Only serious adverse events (SAEs) were assessed. There were no SAEs reported during the conduct of this study.
Arm/Group | Participants With Parkinson's Disease
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.